CLINICAL TRIAL: NCT04546685
Title: Efficacy of a 1-Session Spanish "Empowered Relief" Videoconference-Delivered Group Intervention for Chronic Pain
Brief Title: Virtual 1-Session Spanish "Empowered Relief" Group Intervention for Chronic Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: SCAN Health Plan (Unknown); The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Beth Darnall, Professor, Stanford University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 74942
Record Dates: First submitted 2020-09-04; First posted 2020-09-14 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Waiting Lists

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (waitlist) (Other): Participants will continue their usual clinical care.
  Interventions: Other: Usual Care
- 1-Session pain relief skills class (online Spanish Empowered Relief) (Experimental): Empowered Relief is a 2-hour one session pain relief skills intervention that is delivered to a group of patients by a Spanish-fluent certified instructor using a standardized treatment manual and electronic slide deck. Content includes completion of a pain survey, pain neuroscience education, information on pain and stress responses, experiential exercises, information on three core pain management skills, completion of a personalized plan for empowered relief, and receipt of a binaural app for daily use.
  Interventions: Behavioral: Empowered Relief

INTERVENTIONS:
Other: Usual Care — Participants who are randomized to the Usual Care group (waitlist for cross-over to ER) will be instructed to continue with their normal pain care. They will receive only study surveys (baseline, 2 weeks, and 1 month). Upon completion of the 1-month study, UC participants will be invited to cross-over and receive ER. Post-class treatment appraisal/satisfaction data only will be collected.
  Other Names: Waitlist
  Arms: Usual Care (waitlist)
Behavioral: Empowered Relief — The participants will attend an online Spanish Empowered Relief class. The two hour group session is delivered by a certified instructor and includes pain neuroscience education, 3 core pain management skills, experiential exercises, completion of a personalized plan for empowered relief. Participants download a Spanish binaural relaxation audio file for daily use.
  Other Names: 1-Session Pain Relief Skills Intervention
  Arms: 1-Session pain relief skills class (online Spanish Empowered Relief)

SUMMARY:
Empowered Relief (ER) is a 1-session pain relief skills intervention that is delivered in-person or online by certified clinicians to groups of patients with acute or chronic pain. Prior work in has shown ER efficacy for reducing chronic pain, pain-related distress, and other symptoms 6 months post-treatment. The purpose of this randomized trial is to conduct the first feasibility and early efficacy test of online Spanish ER delivered to Spanish-speaking adult patients with chronic pain. Participants will be followed for 1 month via 3 follow-up surveys (immediately after treatment, 2 weeks and 1 month post-treatment).

DETAILED DESCRIPTION:
Poor access to behavioral pain care contributes substantially to chronic pain burden, particularly for underserved populations such as non-English speaking patients. Empowered Relief (ER) is an evidence-based 1-session (two hour) intervention that rapidly equips individuals with effective pain relief skills. Published evidence from four randomized trials suggest benefits in pain and symptom reduction up to 6 months later. While Spanish ER is being delivered by certified instructors in the U.S., Chile, Spain, Mexico and Puerto Rico, no study has examined patient perceptions and early treatment outcomes for Spanish ER. The investigators will conduct a randomized feasibility and short-term efficacy trial in 110 Spanish speaking patients with chronic pain. The investigators will compare online Spanish Empowered Relief® (ER) vs. Usual Care (UC) in patients with chronic pain of any type (>= 3 months). Participants will be 1:1 randomized to either ER or UC. The study primary endpoint is change in pain intensity or pain interference from baseline to 1 month follow-up (short-term efficacy). UC will be invited to cross over to ER after their 1-month survey (treatment appraisal and satisfaction data only will be collected after receipt of ER).

Aim 1: Test the feasibility of online group-based Spanish ER. Hypothesis 1a: Outcome 1, participant ratings will be >80% for the 7-item treatment appraisal/satisfaction measure administered immediately after completion of ER.

Hypothesis 1b: Outcome 2, ER attendance will be >70%.

Aim 2 (preliminary efficacy): Compare ER vs. UC for reducing multi-primary outcomes (pain intensity or pain interference) and secondary outcomes at 1 month post-treatment.

Hypothesis 2a: Outcome 3, ER will be superior to UC for reducing pain intensity or pain interference from baseline to 1 month follow-up (multi-primary study endpoint).

Hypothesis 2b: Outcome 4, ER will be superior to UC for reducing 4 priority secondary outcomes (sleep disturbance, pain catastrophizing, pain bothersomeness, and anxiety) from baseline to 1 month follow-up.

Hypothesis 2c: Outcome 5, ER will be superior to UC for reducing other secondary outcomes (satisfaction with social roles and responsibilities, anger, fatigue, pain self-efficacy, and depression) from baseline to 1 month follow-up. Patient outcomes will be longitudinally tracked at week 2 and 1 month after the intervention session for ER participants, and at week 2 and 1 month for the UC group.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18+
2. Chronic pain (at least 3 months or more)
3. Spanish fluency
4. Ability to adhere to and complete study procedures

Exclusion Criteria:

1. Cognitive impairment
2. Previous participation in the Empowered Relief class

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-06-12 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Treatment appraisal | Immediately post-treatment
  7 items assess treatment appraisal/satisfaction using 7-point scales (0-6) where higher ratings represent greater appraisal/satisfaction with the treatment. The investigators hypothesize >=80% ratings for treatment appraisal/satisfaction rated immediately post-treatment.
Class Attendance | At treatment
  At least 70% attendance for the registered Empowered Relief online class cohorts.

SECONDARY OUTCOMES:
Pain intensity | Post-treatment 1-month
  Pain intensity: within-subject baseline to 1 month using the Patient Reported Outcomes Measurement Information Systems (PROMIS) Pain Intensity 1-item scale assesses average pain intensity for the past 7 days (0= "No pain" to 10= "Worst pain imaginable") where a higher score represents a greater degree of pain intensity.
Pain interference | Post-treatment 1-month
  Pain interference: within-subject baseline to 1 month using the Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference 8-item scale assesses pain interference with life enjoyment, concentration, and daily activities over the past 7 days. Responses range from 1 = "Not at all" to 5 = "Very much" where higher scores represent a greater degree of pain interference.
Sleep disturbance | Post-treatment 1-month
  Sleep disturbance: Within-subject baseline to 1 month using the Patient-reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance 6-item scale assesses sleep quality over the past 7 days. Responses range from 1 to 5 where higher scores represent lower sleep quality.
Pain catastrophizing | Post-treatment 1-month
  Pain Catastrophizing: Within-subject baseline to 1 month, the Pain Catastrophizing 13-item scale quantifies an individual's pain experience. Scores range from 0-52 with higher scores indicating higher levels of pain catastrophizing.
Pain bothersomeness | Post-treatment 1-month
  Pain bothersomeness: Within-subject baseline to 1 month the Pain Bothersomeness 1-item scale rated 0-10 assesses pain bothersomeness over the past 7 days. Higher scores represent a greater degree of pain bothersomeness.
Anxiety | Post-treatment 1-month
  Anxiety: Within-subject baseline to 1 month the Patient Reported Outcomes Measurement Information System (PROMIS) Anxiety 6-item scale assesses fearfulness, worry and nervousness in the past 7 days. Responses range from 1 = "Never" to 5 = "Always" where higher scores represent greater degree of anxiety.
Satisfaction with participation in social roles | Post-treatment 1-month
  Satisfaction with participation in social roles: Within-subject baseline to 1 month the PROMIS Satisfaction with Participation in Social Roles 7-item scale assesses satisfaction with performing one's usual social roles and activities. Responses range from 1 = "Not at all" to 5 "Very much" where higher scores represent greater satisfaction.
Anger | Post-treatment 1-month
  Anger: Within-subject baseline to 1 month the Patient Reported Outcomes Measurement Information System (PROMIS) Anger 5-item scale assesses anger over the past 7 days. Responses range from 1 = "Never" to 5 = "Always" where higher scores represent a greater degree of anger.
Fatigue | Post-treatment 1-month
  Fatigue: Within-subject baseline to 1 month the Patient Reported Outcomes Measurement Information System (PROMIS) Fatigue 8-item scale assesses fatigue over the past 7 days. Responses range from 1 = "Not at all" and "Never" to 5 = "Very much" and "Always" where higher scores represent a greater degree of fatigue.
Depression | Post-treatment 1-month
  Depression: Within-subject baseline to 1 month with the Patient Reported Outcomes Measurement Information System (PROMIS) Depression 6-item scale assesses negative mood in the past 7 days. Responses range from 1 = "Never" to 5 = "Always" where higher scores represent greater degree of depression.
Pain Self-Efficacy | Post-treatment 1-month
  Pain Self-Efficacy: Within-subject baseline to 1 month with the Pain Self-Efficacy 2-item scale assessing confidence in functioning in the presence of pain. Responses range from 0 = "Not at all confident" to 6 = "Completely confident" where higher scores represent greater confidence in functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Beth Darnall, PhD, Principal Investigator — Stanford University
Locations (1):
- 1070 Arastradero Rd, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ziadni MS, Gonzalez-Castro L, Anderson S, Krishnamurthy P, Darnall BD. Efficacy of a Single-Session "Empowered Relief" Zoom-Delivered Group Intervention for Chronic Pain: Randomized Controlled Trial Conducted During the COVID-19 Pandemic. J Med Internet Res. 2021 Sep 10;23(9):e29672. doi: 10.2196/29672. PMID 34505832
- [Derived] Ziadni MS, Anderson SR, Gonzalez-Castro L, Darnall BD. Comparative efficacy of a single-session "Empowered Relief" videoconference-delivered group intervention for chronic pain: study protocol for a randomized controlled trial. Trials. 2021 May 22;22(1):358. doi: 10.1186/s13063-021-05303-8. PMID 34022930